CLINICAL TRIAL: NCT06743542
Title: Assessment of Handwriting Skills in a Sample of Egyptian Children with Attention-Deficit Hyperactivity Disorder
Acronym: ADHD
Status: Completed | Type: Observational
Sponsor: October 6 University (Other)
Collaborators: National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Walid Saber Hussain, DR, October 6 University
Other Study IDs: o6u; Assessment of Handwriting Skil (Other: O6U)
Record Dates: First submitted 2024-10-25; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Attention Deficit Disorder with Hyperactivity (ADHD)
Keywords: ADHD; Handwriting skills
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | US Export: No

SUMMARY:
PURPOSE: To assess handwriting difficulties in ADHD children. BACKGROUND: Attention deficit hyperactivity disorder (ADHD) is one of the most common neurodevelopmental disorders that affects 7.6% of children worldwide. In addition to the core symptoms defining Attention-Deficit/Hyperactivity Disorder (ADHD), ADHD children often experience motor problems, including graphomotor movements, leading to handwriting difficulties. Studies have confirmed that handwriting skills are adversely impacted by the presence of ADHD, and this is associated with lower academic achievement and self-esteem. Children with ADHD have been found to display greater difficulties in the development of motor coordination, especially in the planning and execution of complex, lengthy, and novel chains of goal-directed behavior. Also, handwriting problems in ADHD may signal underlying executive function deficits such as inhibition, emotional dysregulation, working memory problems, and difficulty with self-monitoring, all of which are required for various daily functions beyond handwriting per se. With a slower motor response and perceptual speed, these deficits may decrease the likelihood that a child with ADHD can work efficiently and stay on-task during school and home activities.

DETAILED DESCRIPTION:
Written informed consents will be obtained from the parents of participants. All participants will undergo the following:

1. Thorough history taking and medical examination.
2. Anthropometric measurements: weight, height
3. Diagnosis by DSM 5
4. Conners' Parent Rating Scales-Revised (CPRS-R) to assess the severity of ADHD symptoms.
5. Intelligence quotient (IQ) test: Stanford Binet intelligence scale, fifth edition to assess the mental ages of the children and measure their intelligence quotients.
6. Assessment of handwriting using (Handwriting Legibility Scale (HLS) to evaluate the handwriting skills of the participants including ……
7. Assessment of neuropsychological abilities related to executive functioning and learning Using the Learning, Executive, and Attention Functioning (Leaf) scale.
8. Language assessment to identify any underlying language deficits that might contribute to handwriting difficulties.
9. A Baseline mechanical gauge was used to measure palmer pinch strength in kilograms
10. A Baseline mechanical gauge was used to measure hand grip strength in kilograms
11. Statistical analysis using the SPSS version 22.

ELIGIBILITY:
Inclusion Criteria:

* ADHD children can read and write
* both sexes.

Exclusion Criteria:

* low IQ children

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ADHD children can read and write both sexes.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Handwriting Skills | 3 monthe

CONTACTS AND LOCATIONS:
Locations (1):
- October 6 university, Giza, Egypt, Egypt